CLINICAL TRIAL: NCT02715362
Title: An Open-label, Uncontrolled, Single-arm Pilot Study to Evaluate Vascular Interventional Therapy Mediated GPC3-targeted Chimeric Antigen Receptor T Cells in Advanced Hepatocellular Carcinoma
Brief Title: A Study of GPC3 Redirected Autologous T Cells for Advanced HCC
Acronym: GPC3-CART
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai GeneChem Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GeneChem GPC3-CART
Record Dates: First submitted 2016-03-11; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: immunotherapy GPC3 CAR-T HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAI-GPC3-CART cells (Experimental): A single dose of GPC3-CART cells will be administered by transcatheter arterial infusion(TAI) mediated as one dose infusion. The dose is 1-10x106/kg GPC3-CAR positive T cells. The infusion will be scheduled to occur 2 days after a single dose of 1.5 grams/m2 of cyclophosphamide. Patients will undergo cannula--DSA radiography--CAR-T cells perfused into hepatic artery. The cells perfusion process would last 15min to 2 h, and the specific time depends on patent's tumor-burdened state.
  Interventions: Drug: TAI-GPC3-CART cells

INTERVENTIONS:
Drug: TAI-GPC3-CART cells — TAI as a local drug delivery pathway, so that more T cells gathered at the tumor site, less T cells to migrated to the normal tissue, thereby enhancing the efficacy of anti-tumor, reducing the potential of side effects. And GPC3-CART is a 2nd CAR, with GPC3 as the target protein, 4-1BB as a co- stimulator
  Other Names: Gene modified patient T cells

SUMMARY:
Intravenous infusion of CART cells in the treatment of solid tumors may be not a suitable choice. Because by intravenous infusion, T cells first entered into the blood circulation, but the number of T cells accumulated at the tumor site is limited, while the probability is high that CART cells contact with normal tissue where target protein is expressed, leading to a more potential off-target side effect. In this study, CART cells infused to the body is mediated by the method of transcatheter arterial infusion(TAI), which is one kind of tumor intervention therapy pathway. We hope by this means could improve the local CAR-T cell numbers，meanwhile reduce the potential side effects.

DETAILED DESCRIPTION:
Patients treated with leukapheresis from which peripheral blood mononuclear cells are purified. T cells are activated and then re-engineered to express chimeric antigen receptors (CARs) specific for GPC3. Cells are expanded in culture and returned to the participant by transcatheter arterial infusion at the dose of .(1-10)×106 CAR positive T cells/kg. The cells perfusion process would last for 15min to 2 h via an ambulatory infusion pump. A single dose of 1.5 grams/m2 of cyclophosphamide will be given two days before CART cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* GPC3 expression positive and histologically confirmed as hepatocellular carcinoma;
* Aged between 18 and 69;
* Persistent cancer after at least one prior standard of care chemotherapy, has no willing for surgery or cannot be suitable for surgery patients;
* Life expectancy greater than 6 months;
* Satisfactory organ and bone marrow function as defined by the following: (1) creatinine <1.5mg/dl; (2) albumin >2; (3) cardiac ejection fraction of >55%; (4) hemoglobin>9g/dl, bilirubin 2.0×the institution normal upper limit;
* Without bleeding disorder or coagulation disorders;
* Dont allergy to Radiocontrast agent;
* Birth control;
* Adequate venous access for apheresis, and no other contraindications for leukapheresis;
* Voluntary informed consent is given.

Exclusion Criteria:

* Pregnant or lactating women;
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary;
* Patients in the situation of: (1) 30 days before apheresis is still in the period of other antitumor drug observation; (2) patient dont recuperate from earlier acute adverse influence brought by any treatments accepted before;
* Four weeks before recruit accepted radiation therapy;
* Previously treatment with any gene therapy products;
* Feasibility assessment during screening demonstrates<30% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation;
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, grade III or IV cardiac disease, serious arrhythmia, liver and kidney disorders or metabolic diseases, CNS diseases);
* Patient with severe acute hypersensitive reaction;
* Taking part in other clinical trials;
* Study leader considers not suitable for this tiral.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-07 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Safety of CAR-T cell infusion mediated by TAI as measured by number of participants with adverse Events | 6 weeks
  To determine the safety and regimen limiting toxicity (RLT) of anti-GPC3 CAR-T transcatheter arterial infusion (TAI) for GPC3-expressing HCC.

SECONDARY OUTCOMES:
Number of participants with tumor response as measured by RECIST | 8 weeks
Detection of CART cells in the circulation using quantitative -PCR | 8 weeks
Serum cytokine levels | 8 weeks
  Measurement of cytokines as indicators of immune response, including IL-2/IL-6/IL-10/TNF/IL-2R

CONTACTS AND LOCATIONS:
Overall Officials: Xu Aimin, Doctor, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided